CLINICAL TRIAL: NCT03185962
Title: Predictors Of Successful Extubation in Critically Ill Patients: Multicentre Observational Study
Acronym: POSE
Status: Completed | Type: Observational
Sponsor: Osaka University (Other)
Responsible Party: Sponsor
Other Study IDs: POSE
Record Dates: First submitted 2017-04-28; First posted 2017-06-14 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Intubation; Extubation; Weaning; Mechanical Ventilation; Liberation From Mechanical Ventilation; Critical Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Successful extubation: extubated successfully
- Extubation failure: reintubated within 48 hours
- NPPV/NHF: use of non-invasive positive pressure ventilation (NPPV) or nasal high flow (NHF) within 48 hours after extubation

SUMMARY:
Extubation failure can directly worsen patient outcomes. Therefore, the decision to extubate is a critical moment during an intensive care unit (ICU) stay. The decision to extubate is usually made after a weaning readiness test involving spontaneous breathing on a T-piece or low levels of ventilatory assistance. However, extubation failure still occurs in 10 to 20% of patients. The investigators focused on previously reported physiological risk factors, and were able to obtain from common clinical practice: 1) age, 2) underlying cardiovascular disease, 3) underlying respiratory disease or occurrence of pneumonia, 4) rapid shallow breathing index (RSBI), 5) positive fluid balance during the previous 24 hours, 6) the ratio of arterial oxygen partial pressure to fractional inspired oxygen, 7) Glasgow Coma Scale, 8) respiratory tract secretions. The investigators aimed to assess the incidence and risk factors for extubation failure among critically ill patients who passed the 30 min spontaneous breathing test (SBT) using a low level of pressure support (PS) with positive end-expiratory pressure (PEEP), in a prospective multicenter study.

DETAILED DESCRIPTION:
Primary Outcome Measures:

Reintubation within 48 hours after extubation (logistic regression will be used to assess the risk factors)

Secondary Outcome Measures:

* Use of non-invasive positive pressure ventilation or nasal high flow within 48 hours after extubation.
* Risk factors for extubation failure, with quantitative variables expressed as means (standard deviation) or medians (interquartiles 25%-75%) and compared using the student t test or Wilcoxon test as appropriate
* Length of ICU and hospital stay, vital status at ICU and hospital discharge, 28-day mortality

ELIGIBILITY:
Inclusion Criteria:

* Mechanically ventilated for longer than 24 hours in Intensive Care Units
* Extubated after successful the 30 min spontaneous breathing test using a low level of pressure support with positive end-expiratory pressure

Exclusion Criteria:

* Decision not to reintubate
* Unplanned extubation
* Extracorporeal circulation
* Patients who died within 48 hours after extubation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients extubated in the ICU
Sampling Method: Probability Sample
Enrollment: 499 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2020-08-25 (Actual)

PRIMARY OUTCOMES:
Implementation of reintubation within 48 hours after extubation | 48 hours
  logistic regression will be used to identify risk factors

SECONDARY OUTCOMES:
Use of non-invasive positive pressure ventilation or nasal high flow within 48 hours after extubation | 48 hours
  logistic regression will be used to identify risk factors
Length of ICU and hospital stay, | 28 days
  mean(standard deviation) or medians (interquartiles 25%-75%) and compared using the student t test or Wilcoxon test as appropriate
vital status at ICU and hospital discharge, 28-day mortality | 28 days
  mean(standard deviation) or medians (interquartiles 25%-75%) and compared using the student t test or Wilcoxon test as appropriate

CONTACTS AND LOCATIONS:
Overall Officials: Yuji Fujino, Study Chair — Department of Anesthesiology and Intensive Care Medicine, Osaka University
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine, Osaka University, Suita, Osaka, Japan

IPD SHARING:
Plan to Share IPD: No